CLINICAL TRIAL: NCT06415097
Title: Benefits of Smart Pens in People With Type 1 Diabetes: a Real-word Retrospective Study.
Brief Title: Benefits of Smart Pens in Type 1 Diabetes
Status: Not yet recruiting | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Francisco Javier Ampudia Blasco, Principal Investigator, Fundación para la Investigación del Hospital Clínico de Valencia
Other Study IDs: SMART PENS_RW
Record Dates: First submitted 2024-01-23; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 1 Diabetes MDI Smart Pen Users: Individuals with type 1 diabetes receiving multiple daily doses of insulin (MDI), utilizing glucose monitoring devices, and using or having used insulin smart pens.
  Interventions: Device: Insulin Smart Pen
- Type 1 Diabetes MDI Smart Pen Non-Users: Patients with type 1 diabetes receiving multiple daily doses of insulin (MDI) and using glucose monitoring devices.

INTERVENTIONS:
Device: Insulin Smart Pen — Retrospective analysis of electronic health records for individuals with type 1 diabetes receiving multiple daily doses of insulin, combined with glucose monitoring devices and who have used or are currently using insulin smart pens.
  Groups: Type 1 Diabetes MDI Smart Pen Users

SUMMARY:
This study aims to address persistent challenges in achieving recommended control goals for patients with type 1 diabetes through innovative interventions. Specifically, the research focuses on assessing the effectiveness of smart insulin pens combined with glucose monitoring devices as a promising treatment option for individuals on multiple daily insulin injections. The study will analyze electronic health records from adults (≥ 18 years) attending the Diabetes Unit of the University Clinical Hospital of Valencia. Participants who are or have used smart insulin pens will be compared with a control group matched for age, sex, duration of diabetes, and HbA1c value at baseline (1:1). Data will be collected on participant characteristics, smart pen usage, glycemic control parameters, and daily insulin doses. The study also aims to identify adverse events associated with the use of smart pens. Ethical considerations include ensuring the anonymity of participant data, and the study is designed to comply with European (EU) data protection regulations. The retrospective nature ensures no interference with physicians' prescription habits.

DETAILED DESCRIPTION:
Rationale:

Despite ongoing advancements in type 1 diabetes management, a significant number of patients continue to struggle in attaining recommended control goals, posing an elevated risk of complications and a diminished quality of life. Hence, there is a need for innovative interventions that genuinely improve diabetes management and associated clinical outcomes. Smart insulin pens, coupled with glucose monitoring devices, emerge as a promising treatment option for individuals on multiple daily insulin injections who may not be suitable candidates for continuous subcutaneous insulin infusion (CSII) therapy. These easy-to-use devices offer significant advantages, such as automated tracking of administered insulin doses along with information other relevant diabetes-related data, facilitating treatment optimization, and helping overcome barriers to achieve better glucose control where both patients and healthcare professionals can implement treatment plans with agility, adopting a more proactive and personalized approach to diabetes care.

While certain recent studies have shown positive outcomes in glycemic control and quality of life linked to the utilization of these devices, there is still a gap in understanding their impact under real-life conditions. Hence, conducting clinical studies within the framework of routine clinical practice becomes imperative to thoroughly assess their application and effects on individuals with type 1 diabetes undergoing multiple daily insulin injections.

The purpose of this study is to provide real-world evidence on the effectiveness of smart pens in enhancing glycemic control and identify specific patient subgroups for targeted interventions.

Hypothesis:

Our hypothesis suggests that the use of smart pens in patients with type 1 diabetes receiving multiple daily insulin doses and utilizing glucose monitoring devices is associated with improved glycemic control. It is expected that the use of these devices is linked to a significant increase in time in range, a reduction in time below the target range, and a decrease in glucose variability during the usage period, compared to a control group.

Primary objectives:

* To describe the clinical characteristics of individuals with type 1 diabetes using smart pens for multiple daily insulin doses in the Valencia Clínico-Malvarrosa Health Department, comparing it with a control group.
* To evaluate changes in glycemic control parameters (HbA1c and continuous glucose monitoring parameters) as well as the incidence of adverse events with the use of smart pens in patients with type 1 diabetes, comparing it with a control group in real-life conditions.

Sample size:

The sample will include all adults (≥ 18 years) with type 1 diabetes who attend or have attended the Diabetes Unit of the University Clinical Hospital of Valencia, using or having used smart insulin pens, along with a control group matched for age, sex, diabetes duration, and HbA1c value at the study's outset (1:1).

Data and study procedure:

Data for this study will be sourced from the electronic health records of adults (≥ 18 years) with type 1 diabetes who attend or have attended the Diabetes Unit of the University Clinical Hospital of Valencia.

The medical records of all participants using or having used smart insulin pens and glucose monitoring devices, as well as a control group (1:1), will be reviewed. Retrospective data will be collected on participant characteristics, the type of smart insulin pen used, and individual changes in glycemic control (HbA1c and glucose monitoring device parameters), as well as daily insulin doses, starting from the date of smart pen prescription. Additionally, all adverse events occurring during the use of smart pens will be documented, specifying their type and frequency for each individual. All data will be compiled in an anonymous Microsoft Excel database, which will be deleted upon completion of the study. Anonymization will be performed by an individual external to the clinical research team.

Ethical aspects:

The study database will not contain any information allowing the individual identification of study participants. The data will be used exclusively for the purposes described in this project. The information will be considered confidential and will be stored and processed in accordance with EU Regulation 2016/679 of the European Parliament and the Council of April 27, 2016, regarding personal data and the free movement of this data, as per Organic Law 3/2018 of December.

Although there are objectives related to medication use, being a retrospective study makes it impossible to alter the prescription habits of any physician in the unit under study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 or above
* Individuals diagnosed with type 1 diabetes
* Individuals receiving multiple daily doses of insulin
* Individuals using a glucose monitoring device
* Individuals who use or have used smart insulin pens since their introduction to the market

Exclusion Criteria:

* Individuals with other types of diabetes
* Individuals utilizing continuous subcutaneous insulin infusion devices
* Individuals using automatic insulin delivery systems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population aged 18 years and older registered in the Population Information System of the Valencian Community (SIP), with an assigned doctor and belonging to the Valencia Clínico - Malvarrosa health department (approximately 320,000 citizens).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Type of smart pen prescribed | up to 24 months
  Type of smart pen prescribed (smart pen prescription)
Type of basal insulin prescribed | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Type of basal insulin prescribed (basal insulin prescription)
Daily dose of basal insulin | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Daily dose of basal insulin (UI/kg)
Number of basal insulin injections | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Number of basal insulin injections per day
Omission of basal insulin | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Omission of basal insulin doses (Yes/No)
Type of prandial insulin prescribed | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Type of insulin prescribed for prandial use (prandial insulin prescription)
Daily dose of prandial insulin | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Daily dose of prandial insulin (UI/kg)
Number of prandial insulin injections | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Number of prandial insulin injections per day
Omission of prandial insulin | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Omission of prandial insulin doses (Yes/No)
Total daily insulin dose | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Total daily insulin dose (UI/kg)
Number of total insulin injections | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Number of total insulin injections per day
Self-monitoring of capillary glucose | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Self-monitoring of capillary blood glucose (SMBG) (Y/N)
Glucose monitoring device | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Glucose monitoring in real-time or intermittently scanned (Yes/No)
Time using the glucose monitoring device | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Percentage of time using the glucose monitoring device
HbA1c concentration | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  HbA1c concentration: at month -3, 0, 3, 6, 12, 18, and 24.
Time in Range (%TIR) | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Time in Range (%TIR): at month -3, 0, 3, 6, 12, 18, and 24.
Time Below Range (%TbR) | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Time Below Range (%TbR): at month -3, 0, 3, 6, 12, 18, and 24.
Time Above Range (%TaR) | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Time Above Range (%TaR): at month -3, 0, 3, 6, 12, 18, and 24.
Mean glucose (mg/dL) | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Mean glucose (mg/dL): at month -3, 0, 3, 6, 12, 18, and 24.
Coefficient of variation of continuous glucose sensor values (CV) | 3 months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  Coefficient of variation of continuous glucose sensor values (CV): at month -3, 0, 3, 6, 12, 18, and 24.
Type of adverse event from the initiation of the prescription of smart insulin pens. | up to 24 months (from the time of the first prescription and throughout the study follow-up)
  Type of adverse event from the initiation of the prescription of smart insulin pens (if any adverse event occurred): severe hypoglycemia, DKA (Diabetic Ketoacidosis), ketosis, other
Months post smart pen prescription when the adverse event occurred. | up to 24 months (from the time of the first prescription and throughout the study follow-up)
  Number of months post smart pen prescription when the adverse event occurred (nº).
Adherence to smart insulin pen usage based on the number of days with data uploads | up to 24 months (from the time of the first prescription and throughout the study follow-up)
  Adherence to data transfer in the mobile application when using the smart pen: at month 6, 12, 18, 24
Smart pen persistence | up to 24 months (from the time of the first prescription and throughout the study follow-up)
  Persistence in the use of smart insulin pens after prescription: at month 6, 12, 18, 24 Persistence defined as the percentage of patients continuing treatment since the first smart pen prescription until discontinuation.
Exclusive use of smart pen | up to 24 months (from the time of the first prescription and throughout the study follow-up)
  Exclusive use of smart insulin pens or mixed use with disposable pens (Yes/No)
Duration of diabetes | up to 12 months
  Duration of diabetes at the time of the first smart pen prescription (years)
Diabetic ketoacidosis | up to 12 months
  Diabetic ketoacidosis (DKA) in the year prior to the initiation of the smart pen (Yes/No)
Severe hypoglycemia | up to 12 months
  Severe hypoglycemia in the year prior to the initiation of the smart pen (Yes/No)
BMI | From three months before the initiation of the first prescription and up to 24 months (throughout the study follow-up)
  BMI (kg/m2): at month -3, 0, 6, 12, 18, 24
Age | up to 12 months
  Age at the time of the first smart pen prescription (years)

CONTACTS AND LOCATIONS:
Overall Officials: F. Javier Ampudia-Blasco, MD, PhD, Principal Investigator — HCUV-INCLIVA
Locations (1):
- INCLIVA, Valencia, Spain